CLINICAL TRIAL: NCT04692350
Title: Adaptation française Des échelles AIDA (Assessment of Identity Development in Adolescence) et LoPF-Q (Levels of Personnality Functioning Questionnaire), Designed to Assess Personality Development in Adolescence.
Brief Title: French Adaptation of the AIDA (Assessment of Identity Development in Adolescence) and LoPF-Q (Levels of Personality Functioning Questionnaire) Scales.
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0621
Record Dates: First submitted 2020-12-30; First posted 2020-12-31 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Personality Disorders; Borderline Personality Disorder
Keywords: Adolescents; Questionnaires
MeSH Terms: conditions — Personality Disorders; Borderline Personality Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — NC
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective of this study is to develop the French version of the two questionnaires AIDA and LoPF-Q. The secondary objective is to investigate the links between disrupted development of identity and adolescent psychopathology.

To participate in the study, patients will have to complete online or paper versions of the questionnaires AIDA-LoPF and other assessments of personality and general psychopathology (BB5, SDQ). Parents will have to answer complete the parent version of the SDQ questionnaire. The BPFSC-11, which is a clinician-rated assessment, will be completed in a subgroup of patients, by the same healthcare professional, in order to assess the concurrent validity. The investigators will also add the clinical diagnoses according to ICD-10 found in the medical record.

DETAILED DESCRIPTION:
A personality disorder is a lasting mode of behavior and lived experience that deviates significantly from what is expected in the culture of the individual is invasive and rigid, appears in early adolescence or adulthood, is stable over time and is a source of distress or impaired functioning.

Most of the tools for assessing high-risk personality disorders and traits have been developed in adults.Yet it is important to have effective tools to distinguish personality disorders from other mental disorders as early as possible. The identification of young people at high risk of personality disorders allows their rapid referral to appropriate psychotherapies.

The AIDA and LoPF-Q, screening questionnaires, were recently developed to include an assessment of personality functioning in the process of diagnosing emotional and behavioral disorders in adolescence. They have been tested in several countries such as Germany, USA, Mexico, Croatia… The results of the studies show that AIDA and LoPF questionnaires are reliable and valid instruments for assessing normal and disturbed identity in adolescents and distinguishes well between patients with psychiatric illnesses and healthy controls.

ELIGIBILITY:
Inclusion criteria:

* The adolescent must be between 12 and 18 years old
* be able (see non-inclusion criteria below) and agree to complete the various evaluations proposed, and not present a psychotic episode at the time. time of the questionnaires.
* The adolescent does not have to have any risky personality traits to participate in this study.

Exclusion criteria:

* insufficient levels of French and / or reading
* presence of an intellectual development disorder or a clinically proven current psychotic disorder,
* active or passive opposition of the patient and / or its legal representatives to participate in the study.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The population studied includes adolescents followed in psychiatry, whether they are hospitalized (UCAP or full hospitalization at MPEA Saint-Eloi in Montpellier) or followed on an outpatient basis (MPEAs Peyre Plantade and Saint-Eloi in Montpellier).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-01-10 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
number of Iinternal consistency | 1 day
  Iinternal consistency (coefficient α) which is supposed to exceed 0.70 at the level of the scale and 0.60 at the level of the subscales.

SECONDARY OUTCOMES:
Number of Inter-item correlational structure (ACP) | 1 day
  Inter-item correlational structure (ACP)
links to psychopathology (especially Borderline personality) | 1 day
  links to psychopathology (especially Borderline personality)

CONTACTS AND LOCATIONS:
Overall Officials: Diane Purper-Ouakil, M.D., Ph. D., Principal Investigator — UH Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC